CLINICAL TRIAL: NCT00773994
Title: Pilot Study Evaluating Characteristic Closure Patterns of the Normal Velopharyngeal Portal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Joseph Losee, Ross H. Musgrave Professor of Pediatric Plastic Surgery Executive Vice-Chair and Program Director Department of Plastic Surgery University of Pittsburgh Medical Center, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07100381
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Cleft Palate
Keywords: anterior palatal eminence; palatal elevation above the maxillary plane; anterior uvular prolapse; "inverted-V" present in base view.
MeSH Terms: conditions — Cleft Palate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Normal velopharyngeal mechanism (Other): All participants in this study are normal healthy adults, who have agreed to undergo to a videofluoroscopic Televex. These participants are acceptable control subjects because they are not diagnosed with VPI and/or submucous cleft palate (SMCP) and the velopharyageal mechanism functions the same in adults as it does in children. This procedure will take approximately 3 minutes to 5 minutes.
  Interventions: Other: Normal Velopharyngeal Mechansim

INTERVENTIONS:
Other: Normal Velopharyngeal Mechansim — The amount of radiation exposure that you will receive from this procedure is about 0.3 rem to the head and neck, with minimal exposure of the other body areas.

SUMMARY:
This prospective research study seeks to determine how the normal velopharyngeal mechanism compares, both anatomically and physiologically, with previous data obtained on subjects with submucous cleft palate (SMCP) in IRB#07080395.

DETAILED DESCRIPTION:
Televex videofluoroscopy utilizes real-time, x-ray imaging to visualize the velopharyngeal port from multiple views or planes. The views generally utilized include the lateral, base and frontal. This technique requires the subject to provide specific speech patterns, as presented by a speech pathologist, while a radiologist obtains adequate views of the velopharyngeal (VP) port. Each procedure will take about 3 to 5 minutes. Fluoroscopic imaging is provided only during speech tasks and swallowing limiting radiation exposure.

1) The radiologist begins by taking a lateral view while speaking, which allows viewing of the velum and posterior pharyngeal wall during speech production, as well as evaluation of cranial base angle, size and location of adenoid tissue, velar length, velar thickness and velar stretch. 2) The speech pathologist gives the subject barium sulfate contrast, approximately 2 to 4 oz, to swallow, which allows for better structure delineation, as well as the confirmation of the presence of palatal fistulae if barium passes through the palate during swallowing. 3) The speech pathologist places the subject in a supine position and barium sulfate is then instilled into the nasal passages bilaterally via syringe, approximately 5 ml. approximately 2. 5 ml in each nostril. This allows for nasopharyngeal coating of structures. 4) The speech pathologist then places the subject in the prone on the table and positioned into a sphinx position with head and neck extended and forearms and palms flat on the fluoroscopic table. The head, shoulders and neck are positioned to find the base view of the velopharyngeal port. This view affords the ability to obtain velopharyngeal closure patterns and size of velopharyngeal defect similar to that of nasopharyngoscopy. 5) The next view obtained by the radiologist is the frontal or anterior-posterior. This is obtained with the head/neck extended to allow for evaluation of the degree of lateral pharyngeal wall motion. 6) The final view obtained by the radiologist is a repeat of the initial lateral view this time with the nasopharyngeal coating in place. This can be beneficial in confirming VPI in the presence of a small VP gap. During the coated lateral view blowing of barium through the VP port can be observed. Additionally if barium is not dissipated during velopharyngeal closure this can be indicative of anatomic VPI. This is all done in the radiology department and takes approximately 3 minutes to 5 minutes.

ELIGIBILITY:
Inclusion Criteria:

* All subjects for this study are adults.
* In this study, the most significant risk is that of radiation exposure, which for Televex videofluoroscopy, is comparable to a single undergoing a single x-ray study, and is significantly less than most CT scans.
* There are no risks to a fetus or pregnant subject involved in this study, nor are there any interventions involved in the research that may be associated with reproductive risks, because all female participants will be given a urine pregnancy test prior to undergoing the Televex Videofluoroscopy.
* All participants will wear protective lead torso and pelvic shields, which are standard for all personnel in a room where a radiologic evaluation is being performed.

Exclusion Criteria:

* The subjects for this study are all adult.
* None of the participants will be children because we are looking for subjects who have reached skeletal maturity which happens around the age of 18 years old
* Any positive urine pregnancy test results would exclude the female subject from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07-15 (Actual)

PRIMARY OUTCOMES:
Normalnormal velopharyngeal mechanism vs abnormal | 2 years or 10 subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Szczepaniak, BS, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States